CLINICAL TRIAL: NCT06903364
Title: Association of Lifestyle With Complications in the Diabetic Population: a Prospective Study
Brief Title: Association of Lifestyle With Complications in the Diabetic Population
Status: Recruiting | Type: Observational
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2025-067
Record Dates: First submitted 2025-03-19; First posted 2025-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group without complications
- Complication group

SUMMARY:
This study is a prospective study of patients with diabetes. The main objective of this study is to investigate the relationship between lifestyle and long-term complications in diabetic patients, which will help to screen out the high-risk group at an early stage and provide scientific advice for the prevention of complications in diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a normative diagnosis of type 2 diabetes
2. Age ≥20 years old, regardless of gender
3. From January 2022 to December 2025, he was treated in Nanfang Hospital

Exclusion Criteria:

1. In the acute infection phase
2. The researchers judged that it was not suitable to participate in this study

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Diabetic patients with or without complications
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Diabetes Complications | From enrollment to the end of the three-year follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- NanFang Hospital of Southern Medical University, Guangzhou, China

IPD SHARING:
Plan to Share IPD: No